CLINICAL TRIAL: NCT05841589
Title: Evaluation of Antimicrobial Efficacy of Green Tea, Garlic With Lime, Pomegranate Extract and Chlorhexidine Mouth Rinses in a Group of Egyptian Children (In-Vivo Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: omnia sayed (Other)
Responsible Party: Sponsor-Investigator, omnia sayed, Principal investigator and demonstrator at Pediatric Dentistry & Dental Public Health Department, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PED18-8M
Record Dates: First submitted 2023-03-27; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Dental Caries
Keywords: herbal mouth rinses; Pomegranate; Caries prevention; Garlic extract; Green tea extract
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: the four groups of the mouth rinses were done in parallel with each other
Who Masked: Participant, Outcomes Assessor
Masking Description: the participant didn't know what he rinsed with the prescribed group of mouth rinse.
  the outcome assessor didn't know what group of mouth rinse belong to the bacterial count that was evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Green tea extract mouth rinse (Experimental): group green tea extract
  Interventions: Procedure: Green tea extract mouth rinse
- Garlic with lime extract mouth rinse (Experimental): garlic with lime extract
  Interventions: Procedure: Garlic with lime extract mouth rinse
- Pomegranate extract mouth rinse (Experimental): pomegranate extract
  Interventions: Procedure: Pomegranate extract mouth rinse
- Chlorhexidine mouth rinse (Experimental): chlorhexidine
  Interventions: Procedure: Chlorhexidine mouth rinse

INTERVENTIONS:
Procedure: Green tea extract mouth rinse — herbal extracts mouth rinse that was prepared in the microbiology laboratory
  Arms: Green tea extract mouth rinse
Procedure: Garlic with lime extract mouth rinse — herbal extracts mouth rinse that was prepared in the microbiology laboratory
  Arms: Garlic with lime extract mouth rinse
Procedure: Pomegranate extract mouth rinse — herbal extracts mouth rinse that was prepared in the microbiology laboratory
  Arms: Pomegranate extract mouth rinse
Procedure: Chlorhexidine mouth rinse — herbal extracts mouth rinse that was prepared in the microbiology laboratory
  Arms: Chlorhexidine mouth rinse

SUMMARY:
the aim of the clinical trial is to evaluate the antimicrobial efficacy of the herbal mouth rinses against chlorhexidine mouth rinse.

DETAILED DESCRIPTION:
The present study was carried out on 84 children. Children were recruited based on certain inclusion criteria after signing a written informed consent by their parents. They were divided into 4 groups. Group (I) the children rinsed with Chlorhexidine mouth rinse, the child rinsed for 1 minute and plaque samples were collected from the child before and after rinsing. Group (II) children rinsed with green tea extract, while group (III) children rinsed with garlic with lime extract and group (IV) the children rinsed with pomegranate extract mouth rinse with the same procedures. .child satisfaction was measured using 5-point pictorial likert scale which is graded from 1 to 5 (1.Excellent.2.Good.3 Average 4.Poor. 5. Very poor).

All the plaque samples were collected and put in sterile test tubes containing thioglycolate as a transport media. They transferred to the microbiology laboratory within half an hour after rinsing for detection of bacterial counts. These samples were incubated 48-96 hours at 37°C. Number of bacterial colonies were counted by hand-held digital colony counter.

ELIGIBILITY:
Inclusion Criteria:• Age 5-8 years.

* No history of systemic disease.
* Patients didn't received antibiotics for at least 3 months before and during the study

Exclusion Criteria:• Children who can't expectorate completely or brush their teeth on their own.

* Fixed or removable orthodontic appliances.
* Children with intra oral abscess, oral lesions or gingival diseases.
* Parental consent was not acquired

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | Through study completion, an average of 1 month
  Child satisfaction was measured using a 5-point pictorial likert scale .This Facial image scale was suitable and easy way to evaluate patient satisfaction about taste, smell and willing to use the mouth rinse. Its format was graded from 1 to 5 while 1 is the most satisfied and 5 is the least satisfied

SECONDARY OUTCOMES:
bacterial count | 1 day after rinsing
  counting of Colony forming units was done by hand- held digital colony counter

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shmas University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No